CLINICAL TRIAL: NCT03922321
Title: A Phase 2a, Multicenter, Open-Label Study of RVT-1401 for the Treatment of Patients With Moderate to Severe Active Graves' Ophthalmopathy
Brief Title: Study of RVT-1401 for the Treatment of Patients With Moderate to Severe Active Graves' Ophthalmopathy (GO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVT-1401-1002
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Graves' Ophthalmopathy
Keywords: IMVT-1401; Graves' Orbitopathy; Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- RVT-1401 (Experimental): RVT-1401 680 milligrams (mg) weekly for two weeks followed by 340 mg weekly for four weeks, administered subcutaneously
  Interventions: Drug: RVT-1401

INTERVENTIONS:
Drug: RVT-1401 — RVT-1401 is a fully human anti-neonatal Fc receptor (FcRn) monoclonal antibody.

SUMMARY:
The purpose of this study was to evaluate safety, tolerability, and pharmacodynamic parameters of RVT-1401 in graves' ophthalmopathy (GO) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Clinical diagnosis of Graves' disease with hyperthyroidism associated with active, moderate to severe GO with a Clinical Activity Score (CAS) ≥ 4 for the most severely affected eye at Screening (on the 7-item scale) and Baseline (on the 10-item scale).
3. Onset of active GO within 9 months of screening.
4. Moderate-to-severe active GO (not sight-threatening but has an appreciable impact on daily life), usually associated with one or more of the following: lid retraction ≥ 2 mm, moderate or severe soft tissue involvement, proptosis ≥ 3 mm above normal for race and gender, and/or inconstant or constant diplopia.
5. Other, more specific inclusion criteria are defined in the protocol

Exclusion Criteria:

1. Use of any steroid (intravenous [IV] or oral) with a cumulative dose equivalent to ≥ 1 g of methylprednisolone for the treatment of GO within 3 weeks prior to Screening.
2. Use of rituximab, tocilizumab, or any monoclonal antibody for immunomodulation within the past 9 months prior to Baseline.
3. Total IgG level < 6g/L at Screening.
4. Absolute neutrophil count <1500 cells/mm3 at Screening.
5. Participants with decreased best corrected visual acuity due to optic neuropathy as defined by a decrease in vision of 2 lines on the Snellen chart, new visual field defect, or color defect secondary to optic nerve involvement within the last 6 months at Screening.
6. Previous orbital irradiation or surgery for GO.
7. Other, more specific exclusion criteria are defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - UBC/VGH Eye Care Center, Vancouver, British Columbia
  - Toronto Retina Institute, North York, Ontario
  - University of Ottwa Eye Institute, Ottawa, Ontario
  - CIUSSS de I'Est-de-I'lle-de-Montreal, Installation Maisonneuve- Rosemont, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 8 participants were screened for the study. Only 7 participants were randomized; 1 participant failed to meet the screening criteria.
Groups:
- RVT-1401: Participants received a RVT-1401 680 milligram (mg) subcutaneous (SC) injection weekly for 2 weeks, followed by a 340 mg SC injection weekly for 4 weeks.
Period: Overall Study
Arm/Group | RVT-1401
Started | 7
Completed | 5
Not Completed | 2
Not completed — Participant Moved | 1
Not completed — Unable to Come to Site Due to COVID 19 | 1

BASELINE CHARACTERISTICS:
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Safety Population: all participants who received at least one dose of study treatment
  Years | 56.7 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Population: all participants who received at least one dose of study treatment
  Participants
    Female | 4
    Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Population: all participants who received at least one dose of study treatment
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 6
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Population: all participants who received at least one dose of study treatment
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 6
    More than one race | 0
    Unknown or Not Reported | 0
Total Immunoglobulin G (IgG), IgG1, IgG2, IgG3, and IgG4 Levels [Mean (Standard Deviation); unit: grams per liter (g/L)] — The serum levels of total IgG and IgG subclasses (1-4) were determined. Population: Pharmacodynamic (PD) Population: all participants who had a Baseline PD measurement and at least 1 post-Baseline PD measurement and received at least 1 dose of study drug
  grams per liter (g/L)
    IgG | 11.29 (1.71)
    IgG1 | 5.11 (1.11)
    IgG2 | 3.74 (0.96)
    IgG3 | 0.61 (0.35)
    IgG4 | 0.49 (0.34)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE), Serious AE (SAE), Treatment-related Adverse Event (AE), and Death During the 6-week Treatment Period
Description: AEs were defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs were defined as AEs that either started on or after the date of the first dose of study drug and on or before the date of the last dose of study drug + 42 days, or had no recorded start date and the stop date was in between the date of the first dose and the last dose of study drug + 42 days. SAEs were defined as any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event that may have jeopardized the participant or may have required medical or surgical intervention to prevent one of the other outcomes listed in the definition.
Time Frame: from Baseline up to Week 6
Population: Safety Population: all participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
Participants
  TEAEs | 7
  SAEs | 0
  Treatment-related AEs | 6
  Deaths | 0

2. Primary Outcome: Number of Participants With Clinically Significant Findings Related to Vital Signs
Description: Clinical significance was determined by the investigator.
Time Frame: up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
Participants | 0

3. Primary Outcome: Number of Participants With a Change From Normal Physical Examination Findings at Baseline to Abnormal Physical Examination Findings at the End of the Study
Description: Abnormality was determined by the investigator.
Time Frame: up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Findings Related to Electrocardiograms (ECGs)
Description: Clinical significance was determined by the investigator.
Time Frame: up to Week 18
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
Participants | 0

5. Primary Outcome: Percent Change From Baseline in Total Immunoglobulin G (IgG), IgG1, IgG2, IgG3, and IgG4 Levels
Description: The serum levels of total IgG and IgG subclasses (1-4) were determined. Percent change from Baseline was calculated as the mean value at the specified time frame (Week 7, Week 6 and 7 combined) minus the Baseline value, divided by the Baseline value x 100. A negative percent change from Baseline represents clinical improvement.
Time Frame: Baseline; Week 7; Week 6 and 7 combined
Population: Pharmacodynamic (PD) Population: all participants who had a Baseline PD measurement and at least 1 post-Baseline PD measurement and received at least 1 dose of study drug. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
Percent change
  Total IgG (Week 6 and 7 combined) | -65.00 (10.78)
  Total IgG (Week 7): number analyzed (Participants) | 3
  Total IgG (Week 7) | -64.83 (17.65)
  IgG1 (Week 7): number analyzed (Participants) | 3
  IgG1 (Week 7) | -67.16 (18.89)
  IgG2 (Week 7): number analyzed (Participants) | 3
  IgG2 (Week 7) | -56.91 (24.66)
  IgG3 (Week 7): number analyzed (Participants) | 3
  IgG3 (Week 7) | -70.05 (21.71)
  IgG4 (Week 7): number analyzed (Participants) | 3
  IgG4 (Week 7) | -61.28 (16.25)

6. Primary Outcome: Mean Change From Baseline in Levels of Anti-thyroid-stimulating Hormone Receptor (Anti-TSHR) Antibodies at Week 7
Description: The serum levels of anti-TSHR antibodies were determined. Change from Baseline was calculated as the Week 7 value minus the Baseline value. A negative change from Baseline represents clinical improvement.
Time Frame: Baseline; Week 7
Population: PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: international units/milliliter (IU/mL)
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
international units/milliliter (IU/mL)
  Baseline | 19.72 (15.073)
  Week 7: number analyzed (Participants) | 3
  Week 7 | -10.59 (9.827)

7. Secondary Outcome: Mean Change From Baseline in Proptosis in the Study Eye and Non-study Eye at Week 7
Description: The study eye was defined as the most severely affected eye at the Baseline visit. In the event that both eyes were affected the same, the right eye was deemed as the study eye. Participants who did not achieve a proptosis response were censored at the date of their last proptosis measurement that occurred in both eyes. Change from Baseline was calculated as the Week 7 value minus the Baseline value. A negative change from Baseline represents clinical improvement.
Time Frame: Baseline; Week 7
Population: PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
millimeter (mm)
  Baseline, study eye | 23.1 (3.34)
  Change from Baseline to Week 7, study eye: number analyzed (Participants) | 4
  Change from Baseline to Week 7, study eye | -1.25 (1.50)
  Baseline, non-study eye | 21.9 (3.63)
  Change from Baseline to Week 7, non-study eye: number analyzed (Participants) | 4
  Change from Baseline to Week 7, non-study eye | -1.25 (0.96)

8. Secondary Outcome: Number of Participants With an Overall Proptosis Response
Description: Proptosis responders were defined as participants with a ≥2 mm reduction in study eye without deterioration (≥2 mm increase) in the fellow eye. Participants who did not achieve a proptosis response were censored at the date of their last proptosis measurement that occurred in both eyes.
Time Frame: Up to Week 18
Population: PD Population
Measure: Count of Participants; unit: Participants
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
Participants | 3

9. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 168 Hours (AUC0-168h) of RVT-1401
Description: Pharmacokinetic (PK) parameters were not estimated because the sparse PK sampling schedule did not allow for accurate estimates of these parameters.
Time Frame: Pre-dose; Day 1, Day 3, Day 5, Day 8, Day 15, Day 22, Day 29, Day 36, Day 38, Day 40, Week 7, Week 8
Population: PK Population: all participants who received at least one dose of study drug and had at least 1 post-dose PK sample assayed for RVT-1401. Only 2 non-Ctrough time point samples were collected after the first dose (on Day 3 and Day 5) and last dose (on Day 38 and Day 40). As a result, having 2 sparse time point samples did not allow to accurately estimate AUC0-168h parameter.
Arm/Group | RVT-1401
Number analyzed (Participants) | 0

10. Secondary Outcome: Maximum Concentration (Cmax) of RVT-1401
Description: PK parameters were not estimated because the sparse PK sampling schedule did not allow for accurate estimates of these parameters.
Time Frame: Pre-dose; Day 1, Day 3, Day 5, Day 8, Day 15, Day 22, Day 29, Day 36, Day 38, Day 40, Week 7, Week 8
Population: PK Population. PK parameters were not estimated because the sparse PK sampling schedule did not allow for accurate estimates of these parameters. Only 2 non-Ctrough time point samples were collected after the first dose (on Day 3 and Day 5) and last dose (on Day 38 and Day 40). As a result, having 2 sparse time point samples did not allow to accurately estimate Cmax parameter.
Arm/Group | RVT-1401
Number analyzed (Participants) | 0

11. Secondary Outcome: Serum Concentration at the End of the Dosing Interval (Ctrough) of RVT-1401
Time Frame: Week 2, Week 3, Week 4, Week 5, Week 6 Day 36, and Week 7
Population: PK Population. Participants with evaluable data were included for the analysis.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
mg/L
  Week 2 | 4.018 (5.9584)
  Week 3 | 12.075 (14.6431)
  Week 4 | 1.284 (2.3063)
  Week 5 | 0.167 (0.1682)
  Week 6 Day 36 | 0.660 (1.5529)
  Week 7: number analyzed (Participants) | 3
  Week 7 | 0.077 (0.0381)

12. Secondary Outcome: Number of Participants With Anti-RVT-1401 Antibody and Confirmed Anti-RVT-1401 Antibody at Week 7
Description: The serum levels of anti-RVT-1401 antibodies were determined. In the initial analysis the samples with responses equal to or above the plate-specific cut-point were identified as potentially positive while those below the cut-point were considered negative. These potentially positive samples were reanalyzed in confirmatory assay. Samples with percent inhibition greater than or equal to the confirmatory cut-point were considered confirmed positive and those below were considered negative.
Time Frame: Week 7
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RVT-1401
Number analyzed (Participants) | 7
Participants
  Initial analysis: negative anti-RVT-1401 antibody | 5
  Initial analysis: potentially positive anti-RVT-1401 antibody | 2
  Confirmed analysis: negative anti-RVT-1401 antibody: number analyzed (Participants) | 2
  Confirmed analysis: negative anti-RVT-1401 antibody | 2

ADVERSE EVENTS:
Time Frame: from Baseline up to Week 18
Description: Treatment-emergent adverse events (TEAEs), defined as AEs that either started on or after the date of the first dose of study drug and on or before the date of the last dose of study drug + 42 days, or had no recorded start date and the stop date was in between the date of the first dose and the last dose of study drug + 42 days, were collected in participants in the Safety Population (comprised of all participants who received at least 1 dose of study treatment) during the treatment period.
Arm/Group | RVT-1401
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RVT-1401 (N=7)
Palpitations (Cardiac disorders) | 1
Lacrimation increased (Eye disorders) | 2
Eye swelling (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Swelling of eyelid (Eye disorders) | 1
Keratopathy (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Superior limbic keratoconjunctivitis (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Weight increased (Investigations) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The PK parameters of AUC0-168h and Cmax were not estimated because of sparse PK sampling schedule.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT03922321/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT03922321/SAP_001.pdf